CLINICAL TRIAL: NCT00303537
Title: Double Blind, Randomized, Placebo Controlled Trial With Metformin in Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Metformin in Non-Alcoholic Fatty Liver Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Aker (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AkerU3
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2007-06

CONDITIONS: Fatty Liver
Keywords: hepatitis; metformin; non-alcoholic fatty liver (NAFLD); non-alcoholic steatohepatitis (NASH); Nonalcoholic fatty liver disease
MeSH Terms: conditions — Fatty Liver; Hepatitis; Non-alcoholic Fatty Liver Disease | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: metformin

SUMMARY:
The study evaluates the use of the antidiabetic medicine metformin in nonalcoholic fatty liver disease.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is a prevalent disorder associated with insulin resistance. Metformin is a drug that has been used for several decades in the treatment of diabetes mellitus. Metformin is known to improve insulin sensitivity. Some authors have reported beneficial effects of metformin in NAFLD, others have not been able to reproduce these findings. Only a few randomized controlled studies have been published so far, and there is still need for controlled trials with sufficient power to assess the efficacy of metformin in this condition.

The aim of this study is to see whether treatment with metformin for 26 weeks results in reduction of liver steatosis (primary endpoint) and reduction in grade of inflammation in those with non-alcoholic steatohepatitis (NASH) (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NAFLD less than 18 months prior to inclusion. For those with pure steatosis, ALAT or aspartate aminotransferase (ASAT) must be elevated above the upper limits of normal, and impaired glucose tolerance or diabetes mellitus type 2 must be present.
* Body weight within +/- 5 kg compared with the weight at the time of biopsy.

Exclusion Criteria:

* Treatment for more than 1 week with metformin or glitazones the last 6 months before inclusion.
* Treatment with insulin.
* Hypersensitivity to metformin.
* Treatment with cimetidine.
* Heart failure requiring pharmacological treatment.
* Coronary heart disease (New York Heart Association [NYHA] class 3 or 4).
* Chronic obstructive lung disease (moderate or severe).
* Breast-feeding or pregnant.
* Metabolic acidosis.
* Renal failure (male [♂]: creatinine > 135 micromol/L, female [♀] > 110 micromol/L).
* Average alcohol consumption > 24 g/day the last year.
* Serum ALAT or serum ASAT > 5 x upper limit of normal (ULN) at screening.
* Cirrhosis.
* Platelets < 100 000.
* Haemochromatosis.
* Alfa-1-antitrypsin-deficiency.
* Wilson's disease.
* Thyroid dysfunction (0.2 mU/L < thyroid stimulating hormone [TSH] < 5.0 mU/L).
* Chronic infection with hepatitis B or C virus or HIV.
* Autoimmune hepatitis (antinuclear antibodies [ANA] > 1/256 or smooth muscle antibodies [SMA] > 1/128).
* Primary biliary cirrhosis (antimitochondrial antibodies [AMA] > 1/64).
* Primary sclerosing cholangitis.
* Previous participation in another clinical trial the last 6 months.
* Legal incapability.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2004-11; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Grade of steatosis as judged by repeat biopsy | 6 mo

SECONDARY OUTCOMES:
Grade of necroinflammation as judged by repeat biopsy | 6 mo
Liver density obtained by computer scan | 6 mo
Serum alanine transaminase (ALAT) | 6 mo

CONTACTS AND LOCATIONS:
Overall Officials: Kaare Birkeland, Prof./Ph.D, Study Chair — Aker University Hospital, Oslo, Norway; Zbigniew Konopski, Cons./Ph.D, Study Chair — Aker University Hospital, Oslo, Norway; Kristian Bjøro, Cons./Ph.D, Study Chair — Rikshospitalet-Radiumhospitalet, Oslo, Norway; John W Haukeland, Physician, Principal Investigator — University Hospital, Aker
Locations (4):
- Norway (4):
  - Haukeland Universitetssykehus, Bergen
  - Aker University Hospital, Oslo
  - Akershus University Hospital, Oslo
  - Universitetssykehuset i Nord-Norge, Tromsø

REFERENCES:
- [Derived] Haukeland JW, Dahl TB, Yndestad A, Gladhaug IP, Loberg EM, Haaland T, Konopski Z, Wium C, Aasheim ET, Johansen OE, Aukrust P, Halvorsen B, Birkeland KI. Fetuin A in nonalcoholic fatty liver disease: in vivo and in vitro studies. Eur J Endocrinol. 2012 Mar;166(3):503-10. doi: 10.1530/EJE-11-0864. Epub 2011 Dec 14. PMID 22170794
- [Derived] Haukeland JW, Konopski Z, Eggesbo HB, von Volkmann HL, Raschpichler G, Bjoro K, Haaland T, Loberg EM, Birkeland K. Metformin in patients with non-alcoholic fatty liver disease: a randomized, controlled trial. Scand J Gastroenterol. 2009;44(7):853-60. doi: 10.1080/00365520902845268. PMID 19811343